## REPUBLIC OF TURKIYE ANKARA YILDIRIM BEYAZIT UNIVERSITY INSTITUTE OF HEALTH SCIENCES

## EVALUATION OF THE EFFECTIVENESS OF VIRTUAL REALITY APPLICATION DURING CESAREAN DELIVERY UNDER SPINAL ANESTHESIA

Data Analysis Plan

**ANKARA-** 30.06.2025

## **Data Analysis Plan**

The data were analyzed using IBM SPSS v23. Normality was assessed using the Kolmogorov-Smirnov and Shapiro-Wilk tests. For the comparison of quantitative variables with normal distribution between two independent groups, the Independent Samples t-test was employed.

For quantitative variables not showing normal distribution between two independent groups, the Mann-Whitney U test was used. The Friedman test was applied to compare three or more related time points. Multiple comparisons were evaluated using the Dunn test.

Associations between categorical variables were analyzed using the Yates correction and the Monte Carlo corrected Fisher's Exact Test. Multiple comparisons among categorical variables were examined using the Bonferroni corrected z-test.

Relationships between non-normally distributed quantitative variables were assessed using Spearman's rho correlation.

Descriptive statistics for quantitative variables were reported as mean  $\pm$  standard deviation or median (minimum–maximum), while categorical variables were reported as frequency and percentage (%).

For advanced analysis, the data were analyzed using Jamovi v2.3.28. The Shapiro-Wilk test was used to assess normality. Robust ANOVA was applied to compare non-normally distributed data across groups and time.

Multiple comparisons were conducted using the Bonferroni test. Quantitative data were presented as median (minimum–maximum). The significance level was set at p < 0.05.

Effect size values were interpreted as follows:  $\leq$ 0.2 indicated a weak effect, between 0.5 and 0.8 indicated a moderate effect, and  $\geq$ 0.8 indicated a strong effect.

The reliability of the scales was evaluated using Cronbach's alpha coefficient. The Cronbach's alpha value ranges from 0 to 1, with values closer to 1 indicating high internal consistency among the items.